CLINICAL TRIAL: NCT06666270
Title: A First-in-human, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Anti-tumor Activity of SYN818, a DNA Polymerase Theta (POLQ) Inhibitor Alone in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of SYN818 for the Treatment of Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou SynRx Therapeutics Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYN-818-101
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Cancer; Metastatic Solid Tumor; Ovarian Cancer; Breast Cancer; Prostate Cancer; BRCA Mutation; HRR Deficiency
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SYN818 tablet (Experimental): SYN818 tablet monotherapy
  Interventions: Drug: SYN818

INTERVENTIONS:
Drug: SYN818 — Patients will orally receive SYN818

SUMMARY:
This interventional study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of SYN818 as monotherapy in adult patients with advanced solid tumors

DETAILED DESCRIPTION:
This study is a Phase I, open-label, multicentre study of SYN818 administered orally in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Having signed the written Informed Consent Form (ICF);
* Male or female aged ≥18 years;
* Life expectancy ≥12 weeks;
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1;
* Patients with histologically or cytologically confirmed locally advanced or metastatic breast cancer, ovarian cancer, prostate cancer or other advanced solid tumors who have experienced disease progression, and available SOC therapies had been exhausted;
* be willing to provide tumor tissue samples (fresh frozen [SF] or previously retained paraffin-embedded [FFPE] tumor tissue samples) or peripheral blood germline DNA or ctDNA sample to detect BRCA mutation, or other deficiency in the HR pathway (by the detection method of next generation sequencing [NGS])
* At least one measurable lesion according to RECIST v1.1;
* No serious hematological, cardiopulmonary, or liver or kidney diseases other than the primary disease;
* Adequate organ function and bone marrow function.

Exclusion Criteria:

* Previous or current use of POLQ inhibitors;
* Hypersensitivity to the active pharmaceutical ingredient or any excipient of SYN818;
* Central nervous system (CNS) metastasis or meningeal metastasis with clinical symptoms, or other evidence indicating that CNS metastasis or meningeal metastasis has not been adequately controlled;
* Other malignant tumors than the study tumors within 5 years prior to the first dose of the study drug, except for localized cancers that have been evidently cured or disease-free for at least 3 years, such as basal or squamous cell skin cancer, superficial bladder cancer, prostate carcinoma in situ, carcinoma in situ of cervix, or carcinoma in situ of breast;
* Patients with Myelodysplastic syndrome (MDS)/Acute myeloid leukemia (AML) or with features suggestive of MDS/AML;
* Dysphagia or refractory nausea and vomiting, malabsorption, extracorporeal biliary shunts, or gastrointestinal disorders that affect drug absorption, e.g., Crohn's disease, ulcerative colitis, or short bowel syndrome, or other malabsorption conditions;
* Major surgery or serious trauma within 4 weeks prior to the first dose of the study treatment or major surgery planned during the trial period, and none of the AEs related to surgery or major trauma have resolved (to ≤ CTCAE v5.0 Grade 1 or baseline level) before the first dose of the study drug;
* History of use within 2 weeks prior to the first dose of the study treatment and need to use protocol-prohibited potent inhibitors or potent inducers of cytochrome P450 (CYP) 3A4/BCRP/P-gp during the study;
* Serious systemic diseases or laboratory abnormalities or other conditions that, at the Investigator's discretion, will make it unsuitable for the patient to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | From first dose of study treatment until the end of Cycle 1 (each cycle is 21-days)
  Severity of adverse events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of participants experiencing adverse events (AEs)/serious adverse events (SAEs) | From time of information consent to 30 days post last dose, up to 3 years
  Number of participants with incidence of adverse events and with serious adverse events including changes from baseline in laboratory parameters, vital signs, ECGs, and physical examination, etc.
Maximum tolerated dose (MTD) | Up to 3 years
  MTD is defined as the maximum dose level at which ≤1 patient have DLTs during the DLT observation period, and it should be determined with 6 evaluable patients.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters and Pharmacodynamic (PD) marker change | Up to 3 years
  Blood drug concentrations at each scheduled time point will be summarized descriptively, and individual and mean concentration-time curves will be plotted by dose group.
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as proportion of patients who achieved complete response (CR) or partial response (PR) according to RECIST 1.1 recorded from first investigational product treatment until disease progression or death due to any cause. The confirmation of response for patients who has PR or CR at first time should be performed by at least 4 weeks. For castration-resistant prostate cancer (CRPC) patients, bone lesion will be assessed according to PCWG3 criteria.
Duration of Response (DoR) and Time to Response (TTR) | Up to 3 years
  DOR is defined, for patients with an objective response, as the time from first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause.
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the time from the first study treatment to the date of the first documentation of objective progression of disease (PD) or death due to any cause.
Serum tumor marker change: CA125, etc. (OC), prostatic specific antigen (PSA, prostate cancer) decreased, and specific tumor markers for other tumor types may also be included (to be assessed by clinical investigators) | Up to 3 years
  The tests for the above serum tumor markers will support the tumor response evaluation.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Fudan University Shanghai Cancer Center., Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No